CLINICAL TRIAL: NCT05931991
Title: Intra-operative Evaluation of the External Ventricular Drain Catheter Position With Structured Light
Brief Title: Intra-operative Evaluation of the External Ventricular Drain Catheter Position With Structured Light for Patients (Bullseye EVD)
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Cari Whyne, Senior scientist, PhD,FIOR, Sunnybrook Health Sciences Centre
Other Study IDs: Bullseye EVD
Record Dates: First submitted 2023-05-31; First posted 2023-07-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Pressure Increase
Keywords: External Ventricular Drain; Intracranial Pressure; EVD malpositioning
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The placement of external ventricular drainage (EVD) is a life-saving procedure used to relieve high pressures in the brain. Often performed at the bedside, a small tube (catheter) is inserted into one ventricle of the brain to drain cerebrospinal fluid and release the pressure build up. In standard practice, EVDs are placed freehand and initial catheter malpositioning occurs in up to ~60% of procedures. Currently, there are no adequate means to verify the position of the catheter before insertion which is a significant impediment to ensure accurate positioning. This non-interventional study aims to validate a novel technology, Bullseye EVD, for verifying the position of the EVD catheter during these emergency procedures.

DETAILED DESCRIPTION:
External ventricular drainage (EVD) is a life-saving procedure used to release cerebrospinal fluid and relieve elevated intracranial pressure due to acute hydrocephalus, often secondary to subarachnoid hemorrhage, spontaneous intracerebral hemorrhage or traumatic brain injury (TBI). To drain cerebrospinal fluid (CSF) from the ventricular system and relieve pressure on the brain, a catheter is inserted into the ipsilateral frontal horn of the lateral ventricle (IFHLV) close to the Foramen of Monro (FoM). Twist-drill trephination is utilized to create a frontal burr hole at Kocher's point, approximately 11.5cm superior to the nasion and 2-3cm lateral of the midline. The dura is perforated, and the catheter is inserted with a rigid stylus. The current standard of care is a freehand technique which is often performed by neurosurgeons at the bedside in the ICU. It relies on surface anatomical landmarks to guide the catheter trajectory towards the FoM perpendicular to the calvarial slope at Kocher's point. However, the freehand technique is challenging to accurately perform, often requiring multiple passes of the catheter through the brain, with trajectory deviation most critical to malpositioning. Up to 24% of malpositioned EVDs require revision or reinsertion which can significantly increase catheter-associated infection. Up to 45.5% of EVD procedures require multiple passes for successful catheter insertion (6). This can lead to hemorrhage along the catheter tract (up to 34%, catheter dysfunction (up to 38%, and catheter-associated infection (up to 36% which increase EVD-associated health care costs (up to 20%). EVD malpositioning outside of the IFHLV (up to 60%) has been associated with other rare but significant complications including coma and diabetes insipidus. Large deviations in catheter placement have resulted in catheter insertion into significant brain regions (thalamus, hypothalamus, basal ganglion, internal capsule. Angular error within the coronal plane is the primary determinant of successful catheter insertion.

Bullseye is a novel intra-procedural system the investigators initially developed for glenoid guidepin placement. Bullseye EVD uses a verification workflow (guess and check) to identify EVD catheter position and trajectory with reference to the diagnostic CT image prior to catheter insertion using structured-light imaging. Structured-light scanning currently has several medical applications due to its speed, accuracy, and robust 3D surface reconstruction, and has been investigated in planning bedside subdural evacuation port system placement. In vitro performance of Bullseye EVD was demonstrated through testing on 3 cadaveric specimens to localize EVD placement on both sides of each of the heads (N=6 trials in total). The success of this in vitro work motivated further development of the technology including clinical evaluation for EVD.

Reducing EVD malpositioning and associated complications is a priority for neurosurgeons, however costly and cumbersome navigation solutions have had limited uptake in this urgent procedure that is often conducted at the bedside. Bullseye EVD represents a portable, safe, low-cost technology that can identify catheter positioning on existing preprocedural CT imaging. The proposed work, including integration into the existing clinical workflow, evaluation of in vivo accuracy and automation to enable rapid feedback during EVD placement, is critical to translating this technology from the bench to the bedside.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Scheduled to undergo placement of an EVD
3. Located in B5 ICU or CRCU
4. Existing pre-procedural head CT imaging

Exclusion Criteria:

1. Set up time poses a safety risk (Clinical discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 15 patients will be enrolled in this study at Sunnybrook Health Sciences Centre's ICU. The PI, study team members who are part of the circle of care, and study personnel will identify potential study participants. The Research Coordinator or assistant will approach for consent.
  Given that the clinical procedure involved- the EVD- is an urgent procedure with short timelines, s deferred consent model may also be used in this study as it satisfies the conditions for deferred consent as set out in the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans - TCPS 2 (2022) Article 3.7A,.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the structured light computer vision system | Data analysis to start immediately post procedure.
  The primary study outcome will be the accuracy of the structured light computer vision system. This will be quantified as the difference between predicted and actual position of the EVD catheter measured as a combined analysis of version error (degrees), inclination error (degrees), and offset error (mm).

SECONDARY OUTCOMES:
Procedural time for Fiducial placement and optical imaging | Time measured during procedure
  The number of minutes required for these additional tasks
Workflow integration | Immediately after procedure
  Analysis of the current workflow and changes required to enable the use of Bullseye EVD
User feedback | Immediately after procedure
  User feedback to evaluate acceptability and utility of the technology by the surgeons and procedural team, and to identify potential barriers and opportunities to improve safe and accurate EVD placement. This will be conducted within a user centred design framework

CONTACTS AND LOCATIONS:
Overall Officials: Cari Whyne, PHD, FIOR, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No